CLINICAL TRIAL: NCT04540380
Title: Renal Allograft Tolerance Through Mixed Chimerism - SMC/MGH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tatsuo Kawai, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tolerance SMC-MGH
Record Dates: First submitted 2020-08-18; First posted 2020-09-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Rituximab; fludarabine; Cyclophosphamide; siplizumab; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rituximab, Fludarabine, Cyclophosphamide, Thymic irradiation and Siplizumab — Conditioning regimen .Patients will receive Rituximab, Fludarabine, Cyclophosphamide, Thymic irradiation and Thymoglobulin
Procedure: Combined bone marrow and kidney transplant — Recipients will receive a conditioning regimen that includes rituximab on study days -7 and -2, fludarabine 10mg/m2/day on days -6 to -3 (4 doses), cyclophosphamide (22.5mg/kg/day) on days -5 and -4, followed by local thymic irradiation (7 Gy) on day -1 and Siplizumabon days -1, 0, and +1. Combined kidney and bone marrow transplant will be performed on study day 0. Methylprednisolone will be started at 250 mg/day on day 0 and tapered to prednisone 20mg by day 10 after which it will be continued until day 20. Prophylaxis will be provided for hemorrhagic cystitis, PCP, fungal infection, CMV, and perioperative infection. All patients who require any blood transfusion will receive only leukocyte-depleted and irradiated blood products for a period of at least 52 weeks following transplantation. The proportion of patients successfully weaned off immunosuppression without chimerism transition syndrome (CTS) will be assessed.

SUMMARY:
The goal is to investigate the safety of the conditioning regimen, and its ability to induce donor/recipient lymphohematopoietic chimerism without Chimerism Transition Syndrome (CTS), which may result in donor-specific unresponsiveness (tolerance) to the renal allograft in the absence of maintenance immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age.
* Candidate for a living-donor renal allograft from an HLA mismatched donor
* Subjects with chronic kidney disease stage or ESRD who are treated with either hemodialysis or peritoneal dialysis.
* First transplant.
* Use of FDA-approved methods of contraception
* Ability to understand and provide informed consent.
* Negative COVID at screening and 2 days before procedure

Exclusion Criteria:

* ABO blood group-incompatible renal allograft.
* Participant with a (non DSA) PRA > 20% within 6 months prior to transplant
* Persistent Leukopenia (WBC less than 2,000/mm3) or thrombocytopenia (<100,000/mm3).
* Seropositivity for HIV-1, hepatitis B core antigen, or hepatitis C virus (confirmed by hepatitis C virus RNA); or positivity for hepatitis B surface antigen.
* Active infection
* Left ventricular ejection fraction < 40% as determined by TTE or clinical evidence of heart failure
* Forced expiratory volume FEV1 or DLCO < 50% of predicted.
* Lactation or pregnancy
* History of cancer (following the American Transplant Society Guidelines)
* Underlying renal disease etiology with a high risk of disease recurrence in the transplanted kidney (such as focal segmental glomerulosclerosis).
* Prior dose-limiting radiation therapy
* Known genetic disease or family history that may result in greater sensitivity to the effects of irradiation, or a physical deformity that would preclude adequate shielding or appropriate dosing during the irradiation component of the conditioning regimen
* Enrollment in other investigational drug studies within 30 days prior to enrollment
* Abnormal (>2 times lab normal) values for (a) liver function chemistries (ALT, AST, AP), (b) bilirubin, (c) coagulation studies (PT, PTT).
* Allergy or sensitivity to any component of Siplizumab, Fludarabine, Cyclophosphamide, tacrolimus, DMSO, MMF or rituximab.
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.
* Subjects who have non-insulin dependent diabetes (NIDDM) without good blood glucose control (HbA1c<7). Subject with severe retinopathy, gastroparesis, or severe neuropathy which prevent subject's normal independent daily activities will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Transient Chimerism | 36 months after immunosuppression withdrawal
Incidence of Chimerism Transition Syndrome | 36 months after immunosuppression withdrawal
Incidence of tolerance induction | 36 months after immunosuppression withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided